CLINICAL TRIAL: NCT02862821
Title: Biomarkers of Online Gambling Addiction: Biomarqueurs de la dépendance Aux Jeux d'Argent en Ligne
Brief Title: Biomarkers of Online Gambling Addiction
Acronym: BLUNDER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: P/2016/292
Record Dates: First submitted 2016-07-20; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Gambling
Keywords: biomarkers of psychiatric disorder; gambling addiction; high resolution-ElectroEncephaloGraphy (HR-EEG)
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- validation of EEfRT task (Experimental): 20 healthy volunteers will be recruted to validate motivation EEfRT task which is adaptated to HR-EEG
  Interventions: Other: HR-EEG
- biomarkers identification (Experimental): 20 addict online poker gamblers and 20 non-addict online poker gamblers will be recruted : After standardized questionnaires to define the socio-demographic data, the diagnosis of gambling addiction (Diagnostic and Statistical Manual of Mental Disorder 5th edition DSM-5), screening for comorbidities addictive, the level of anxiety and impulsivity, brain acvtivity will be registred (by randomisation between the 2 tasks) with HR-EEG: during the performance of a task of motivation evaluation laboratory (EEfRT) adaptated for high-resolution electroencephalography AND during a laboratory task that assesses decision making in conditions of uncertainty (IGT) with its version for high-resolution electroencephalography has already been validated in a previous study (Giustiniani et al., 2015).
  Interventions: Other: HR-EEG
- biomarkers validation (Experimental): 13 online poker gamblers will be recruted, independently of their dependance profile and they will realize the same task that in precedent arm (quaestionnaires and 2 tasks adaptated to HR-EEG).
  Interventions: Other: HR-EEG

INTERVENTIONS:
Other: HR-EEG

SUMMARY:
The purpose of this study is to identify alterations of motivational processes related to decision making in uncertainty condition associated with gambling addiction: by studying the dynamics between brain systems involved in decision making and motivation.

DETAILED DESCRIPTION:
Internet gaming is a major risk for the vulnerable in terms of risk of dependence, emergence of psychiatric disorders, financial consequences, and family. Addictions to games in France represent 1 to 2% of the general population. Online poker happens to be a specific form of gambling which has the fastest growing online games. If vulnerabilities factors have been reported in many studies, to date no biomarkers for screening people at risk are available.

One of the favorite way in biomarker research concern impaired decision-making capacity biomarkers. In a previous work, investigators have shown that the decision was strongly linked to motivation and impaired decision-making capacity would be associated with a motivational dys-regulation (Giustiniani et al., 2015) .

The search for biomarkers in parallel to the motivation of the decision making is essential and yet this day nonexistent in the literature. Here, with subjects addicted to online poker, a behavioral protocol developed to measure motivation in pathological populations (Effort-Expenditure for Rewards Task, EEfRT) will be used and will be specifically adapted to be studied by functional neuroimaging.

The main objective is to identify alterations of motivational processes related to decision making in conditions of uncertainty associated with gambling addiction. For this purpose, the dynamics between brain systems involved in decision making and motivation will be studied.

As a secondary objective, correlations between neural activity and performance to different tests used to measure decision making (Iowa Gambling Task IGT) and motivation (EEfRT) will be evaluated. Finally the influence of motivation level on the performance score to decision making task will be evaluated, the goal will be the development of an optimal strategy in terms of prevention.

The study will be conducted at the University Hospital of Besancon during 36 months with 73 participants:

The experiment will involve three stages:

* stage 1 : validation of HR-EEG adaptated motivation EEfRT task adaptated to HR-EEG by 20 healthy volunteers .
* stage 2: identification of biomarkers by 20 addict online poker gamblers and 20 non-addict online poker gamblers
* stage 3 : validation of previously identified biomarkers by 13 online poker gamblers recruted in poker forum.

All stages progress according to the same plan:

* Standardized questionnaire to define the socio-demographic data, the diagnosis of gambling addiction (ICJE criteria (Indice Canadien fu Jeu Excessif), screening for comorbidities addictive, the level of anxiety and impulsivity.
* Registration of brain activity (randomisation): during the performance of a task of motivation evaluation laboratory (EEfRT) adaptated for high-resolution electroencephalography AND during a laboratory task that assesses decision making in conditions of uncertainty (IGT) with its version for high-resolution electroencephalography has already been validated in a previous study (Giustiniani et al., 2015).

Statistical analysis will aim to compare the average activation differences between the two populations for each functional neuroimaging examination. Then a subject-by-subject analysis of each brain activation will be conducted to look for correlations between the various examinations and strength of neuronal response.

Following this study, the results will allow us to identify biomarkers of addiction that will help improving vulnerable populations screening capabilities to tailor prevention strategies. Furthermore the identification of specific neural correlates dependence will adapt therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* stage 1: healthy volunteers (no online poker gamblers and no-addict (excepted tobacco and caffeine))
* stage 2 : 20 addict-online pokers gamblers and 20 non addict online pokers gamblers (according to ICJE criteria)
* stage 3 : 13 online poker gamblers (independently of their dependence level)

Exclusion Criteria:

* left-handed
* female
* stage 1 and 2: other addictive pathology excepted tobacco and caffeine

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
average activation for each functional neuroimaging examination | day 7 ; day 14

SECONDARY OUTCOMES:
correlations between various examinations and strength of neuronal response | day 7 ; day 14
  a subject-by-subject analysis of each brain activation will be conducted to look for correlations between the various examinations and strength of neuronal response.

CONTACTS AND LOCATIONS:
Overall Officials: Julie GIUSTINIANI, MD, Principal Investigator — University Hospital of Besancon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giustiniani J, Gabriel D, Nicolier M, Monnin J, Haffen E. Neural Correlates of Successful and Unsuccessful Strategical Mechanisms Involved in Uncertain Decision-Making. PLoS One. 2015 Jun 18;10(6):e0130871. doi: 10.1371/journal.pone.0130871. eCollection 2015. PMID 26086196